CLINICAL TRIAL: NCT05566977
Title: Autologous Adoptive T Regulatory Cell Transfer in Autoimmune Diseases: Anon-randomized Open Label Phase 1 Pilot Study
Brief Title: Autologous Adoptive T Regulatory Cell Transfer in Autoimmune Diseases.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, zeinab ahmed yousif hasan ashour, professor of internal medicine, allergy and clinical immunology, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMASU P19a/2022
Record Dates: First submitted 2022-09-21; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Lupus Nephritis; Type 1 Diabetes Mellitus
Keywords: T regulatory cells ,lupus nephritis ,type 1 diabetes .
MeSH Terms: conditions — Lupus Nephritis; Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: refractory lupus nephritis type one diabetes in adults
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with autoimmune disease :lupus nephritis and type1 diabetes melitus (Experimental): single arm of patients with autoimmune diseases : patients of the first group selected as refractory lupus nephritis. patients of the second group of autoimmune diseases are selected to have type1 diabetes Meletus.
  Interventions: Other: autologous adoptive T regulatory cell transfer.

INTERVENTIONS:
Other: autologous adoptive T regulatory cell transfer. — Identification and count, using flowcytometry, for human Tregs will be based on both positive and negative cell markers, human Tregs are (CD4+, CD25+, CD127-, Foxp3+). Peripheral heparinized venous blood will be used .GMP-Compliant Protocol for the Isolation and Expansion of Tregs for Clinical Application .Cryopreservation of Expanded Tregs .Administration of T reg cells and follow-up of adverse events.

SUMMARY:
Investigators aim to develop an effective and safe treatment of autoimmune diseases through adoptive T regulatory cells transfer. Our objectives are to evaluate the safety and efficacy of autologous adoptive Treg (CD4CD25FoxP3 CD127 low regulatory) cell transfer to patients with refractory autoimmune diseases: Refractory lupus Nephritis, and adults' type1 diabetes mellitus. Patients and Methods: This is Non randomized open label phase 1 pilot study including ten patients with refractory lupus nephritis and ten patients with Type 1 diabetic patients. All patients will be subjected to Full history taking, clinical examination and pretreatment investigations according to the type of autoimmune disease then regulatory T cells (Tregs) identification and count, Treg isolation and expansion and finally administration of T reg cells and follow-up of adverse events and outcomes.

DETAILED DESCRIPTION:
Autoimmune disorders are chronic diseases caused by the breakdown of tolerance against self-antigens

; one hypothesis involves a failure in central and peripheral tolerance with the latter being associated with reduced Treg (CD4+CD25+FpxP3CD127- T- Regulatory )cells number or failure in their function (6).

In preclinical studies, human CD4+CD25+CD127- Treg cells have been shown to be effective in preventing Graft vs. Host Disease (GvHD) (7, 23), autoimmune diseases (13,22) and delaying graft rejection (19, 26).

The positive outcomes gave the rationale to apply Treg cells for the treatment of human diseases and results from the first clinical trials with adoptively transferred Treg cells investigators published in 2009 (24).

What does this study add? This is the first interventional study on adoptive Treg cell transfer in Egypt as a therapeutic trial for patients with refractory autoimmune diseases who do not respond to base line of care treatment available in the institute. Separation of this Treg cells was done in Egyptian patients but as a descriptive study only (as mentioned below).

investigators choose two diseases in order to give some chance for success for getting fund of our research, as its cost is expensive. Investigators chose these two diseases (refractory lupus nephritis and type 1 diabetes in adults, as they are the commonest trials in international publication).

investigators will evaluate the safety and efficacy of autologous adoptive Treg(CD4CD25FoxP3 CD127 low regulatory) cell transfer to patients with refractory autoimmune diseases: Refractory lupus Nephritis and adults type1 diabetes mellitus.

2.STUDY QUESTION/AIM / OBJECTIVES investigators will evaluate the safety and efficacy of autologous adoptive Treg (CD4CD25FoxP3 CD127low regulatory ) cell transfer to SLE patients with refractory lupus nephritis and patients with adult type1 diabetes mellitus.

Monitoring plan of AE is documented in the protocol checking for systemic and local adverse events using CTCAE(5).Safety assessments will consist of continuous monitoring and reporting of adverse events (AEs) (with monthly visits or as clinically indicated by mobile contact or out patients visits); monitoring of vital signs, , physical examinations and laboratory assessments. Precise documentation and proper management will be done for any AE that may occur (in the outpatient and inpatient units as indicated).Patients will be seen monthly for detection of any adverse event or as clinically evaluated by Mobil contact The following will be assessed:

1. White blood cell count (WBC) with differential count , red blood cell count (RBC), platelet count (PLT), hemoglobin (Hb) and hematocrit (Hct).
2. Liver functions, kidney functions tests and electrolytes measurement.

   Efficacy of adoptive Treg cell transfer:
   * Clinical Evaluation: Full history taking and thorough clinical examination with assessment of disease activity score (clinically and laboratory) to compare with baseline data.
   * Laboratory testing according to the type autoimmune disease:

     1. Laboratory tests for detection of disease exacerbation,
     2. CD4CD25FoxP3,CD127low cell count in peripheral blood sample ,
     3. Serum cytokine detection (INF-gama,TNF-alpha,IL1,IL2,TGF-beta,IL-10,IL-17)
   * Radiological evaluation if needed according to the type of autoimmune disease:

     1. Ultrasound
     2. CT scan
   * Researchers will detect the efficacy of T reg cells infusion after 3 months, after 6 months and after one year of administration.
3. METHODOLOGY:

Type of Study : Non randomized open label phase 1 pilot study Study Setting: Table of responsibilities (Table 1) :see below Study duration: Two years.

Study Population:

* Ten Systemic lupus erythematosus (SLE) patients with refractory lupus nephritis: inclusion and exclusion criteria
* Ten Type 1 diabetic patients: inclusion and exclusion criteria

Sampling Method:

Purposive samples following pre-set inclusion and exclusion criteria.

Sample Size:

Researchers will include ten patients in each autoimmune disease as a pilot study.

Study Procedures:

* First Visit: Rheumatology team and Endocrinology team will select patients according to the above-mentioned criteria from internal medicine department of ASU Hospitals. Full laboratory and Immunological investigations will be done in ASU Hospital central labs. Nurses in medical out patient's clinic of ASU Hospitals will withdraw the blood samples from all cases. Patients will do all required imaging modalities in the Radio diagnosis department, ASU Hospital. Rheumatology team and Endocrinology team will take a written consent from all patients included in the study.
* Second visit: After the first visit by one week. Patient will come to internal medicine department. All Patients will be evaluated clinically, laboratory, and radiological as indicated for detection of severity or activity of the disease. Patient will go to the medical research Centre for peripheral blood sampling under sterile conditions for separation of Treg cells. The distance between the research Centre and medical departments is around 200 m .The hospital transferring car will transfer patient (golf car) for 150 m after walking for 50 m.
* Third visit: (after the second visit by six weeks):patient will come to the medical research Centre for Admission under supervision of Allergy and immunology team for administration of T reg cell infusion. Allergy and Immunology team will follow up patient for 24 hours after infusion.
* Detection of adverse events will be checked monthly. Mobile contact between patient and both rheumatology, endocrinology and clinical immunology teams will be kept for recording any adverse event.
* Fourth Visit: (after three months of third visit):Medical team will do full laboratory, immunological and radiological follow up in ASU central lab and ASU radiology department after three months of T reg infusion. Clinical scoring and detection of activity and severity of the disease will be recorded.
* Fifth Visit after six months of infusion. The same will be done as visit 4.
* Final visit after one year for detection of any adverse event.
* Ethical committee will be informed by a full report including all clinical and laboratory data about the last six steps for each patient who received the t reg cell infusion as recorded by immunology rheumatology and endocrinology teams. Figure 2 shows scheme for procedures and follow up.

All Patients will be subjected to the following:

In the first visit

* Full history taking and clinical examination including assessment of the severity and clinical disease activity scoring according to the type of autoimmune disease.
* Pretreatment investigations CBC with differential WBCS count , total lymphocytes, red blood cell count (RBC), platelet count (PLT), hemoglobin (Hb) and hematocrit (Hct)
* liver functions, kidney function tests and electrolytes (Na, K, and Ca)evaluation.
* Liver function tests: serum albumin ,PT and INR .bilirubin total and direct .AST ,ALT, Alkaline phosphatase ,Serum albumin.
* Kidney function tests (serum creatinine ,BUN )and electrolytes ( serum Na ,K and, Ca)
* ESR and CRP.
* Evaluation of CD4+CD25+FoxP3+CD127- cell count before intervention, after three months and after 6 months of the intervention by flowcytometery.
* Serology tests for all patients: INF- gamma, TNF -alpha, IL-17, IL-2, IL-10, and TGF-beta. All cytokines will be done by ELISA test before adoptive T reg transfusion, after 3 months and after 6 months of transfusion.
* Radiology investigations according to the type of autoimmune disease and if indicated.
* Laboratory tests according to the autoimmune disease:

SLE patients:

* Fasting and 2-h postprandial blood glucose, complete blood count (CBC), complete urine analysis,
* Measurement of proteins in 24 h urine (g/24 h).
* Antinuclear antibodies (ANA) titer and pattern and anti-double stranded DNA antibodies (anti-dsDNA measurement will be done by immunofluorescence technique, where titer of 1/40 or more is considered positive)
* Serum complement level (C3 and C4).

T1D Patients:

* Fasting C-peptide levels,
* fasting glucose, HbA1c and
* T1D autoantibody [glutamic acid decarboxylase autoantibody (anti-GAD65), insulin autoantibody (IAA), insulin antigen 2 antibody (IA2) or zinc transporter 8 autoantibody (anti-ZnT8)] levels will be measured.

Regarding blood samples: our plan as regards frequency and amount of blood samples as following:

A- Frequency:

* Base line for CBC, KFT, LFT, electrolytes, after 3 months and after 6 months of intervention.
* Detection of T reg count before infusion ,after three months and after 6 months
* In case of grade 2 or more adverse events.

B- Amount:

* For base line evaluation and preparation: 6 ml (2ml * 3 tubes). The same amount after 3 months and after six months of T reg infusion.
* Detection of T reg count: 4 ml (2ml* 2 tubes) for hematology and chemistry.
* Separation of T reg Cells For culture and expansion: ( 400ml )
* In case of adverse events: as clinically indicated, from 2 ml to 4 ml. Regulatory T cells (Tregs) identification and count(10) Identification and count, using flowcytometry, for human Tregs will be based on both positive and negative cell markers, human Tregs are (CD4+, CD25+, CD127-, Foxp3+).

Cryopreservation of Expanded Tregs:

In order to allow infusion of the cell product several times, the feasibility of Treg cryopreservation will be used. Cryopreservation of Tregs allows flexibility in administration to assist with clinical pathways and facilitates completion of all required release assays. ( 10 ) Administration of T reg cells and follow-up of adverse events Results of blood chemistries and hematology will be reviewed, and a history of any recent illness or fever will be obtained before infusion of the cells. Patients will receive premedication with paracetamol and diphenhydramine. Poly t regs will be infused via a peripheral intravenous line over 10 to 30 min.

Vital signs will be taken before and after infusion, then every 15 min for at least 1 hour, then every hour for the first 4 hours, and every 4 hours for 20 hours. Chemistries and complete blood count with differential blood count will be repeated the next day before discharge from the clinical research unit. Patients will be seen for follow-up assessments on day 4 after infusion, then weekly for 4 weeks, then after 13weeks, and then after 26 weeks. Telephone monitoring for adverse events will continue one year after infusion followed by a final clinic visit.

The dose of ex-vivo expanded T reg will be the same for all patients. It will be administered in increasing doses of 5x10^6-1x10^8 cells I V infusion I V infusion. It is the minimum dose in previous international therapeutic cohorts in order to achieve safety (14).

ETHICAL CONSIDERATIONS

1. RISKS and MINIMIZATION OF RISKS:

   * Possible Risks of Ultrasound Medical Imaging: Ultrasound medical imaging is a fast and safe way to evaluate patients that do not represent any risk and do not lead to side effects. They do not lead to any change in the patient's original condition, but there may be rare problems such as: pain or bruising.
   * Complications of venipuncture: hematoma formation, nerve damage, pain, hemoconcentration, extravasation, iatrogenic anemia, arterial puncture, petechiae, infection, syncope and fainting, excessive bleeding, edema and thrombus. To minimize these risks it will be taken under aseptic conditions by qualified nurses.
   * Risk of infection: T reg cell isolation and expansion will be done under strict sterilized environment. Frequent sterility techniques will be followed during expansion and Quality control, and release assays will be done before adoptive T cell transfer.

     ● Side effects of taking 400 cc of blood from patients: like that of blood donation which are rare and include the development of a local traumatic hematoma when the needle is removed from the vein. Holding local pressure and application of ice or cold compresses to the area can help to prevent the development or progression of hematomas. These hematomas are usually small and do not cause major problems. Development of dizziness, sweating and syncope might also occur, and can be avoided by requiring the patient to sit in a reclined position for a few minutes, and when able, slowly moving to the upright position and moving to an area where they will be given something to eat and drink. Increased fluid intake will be encouraged over the few hours following taking the blood. Patient Hb level must be not less than 11g/dl before withdrawal of blood for Treg isolation. investigators will prepare packed RBCs before blood withdrawal in order to be given if indicated clinically.
   * Risk of infection / inflammation: Treg cell isolation and expansion will be done under strict sterilized environment. Frequent sterility techniques will be followed during expansion and Quality control, and release assays will be done before adoptive T cell transfer .The accepted release criteria include: Phenotype>60%, , viability :> 70%, sterility and negative mycoplasma.
2. DISCONTINUATION CRITERIA (STUDY AND ENROLLMENT TERMINATION) Safety Stopping Rules for Individual Subjects

   Treatment will be discontinued in any subject who experiences any one of the following:
   * Any SAE, or a clinically significant grade 4 AE or confirmed grade 4 laboratory abnormality for an individual subject, which is considered by the investigator to have a reasonable possibility of relatedness to T reg infusion. Subjective clinical symptoms not reflecting major organ dysfunction, such as severe headache, may or may not warrant treatment discontinuation in the judgement of the investigator.
   * Subjects may voluntarily discontinue treatment or withdraw from the study at any time.
   * They may also be removed from the study at any time if the investigator determines that continuing the study would result in a significant safety risk to the subject.
   * Persistent noncompliance with the protocol requirements Subjects who prematurely discontinue study treatment should be encouraged to maintain the same protocol schedule and assessments as described for continued follow-up for key study outcome data.

   Study Stopping Rules

   This clinical trial will be paused for any of the following reasons:
   * Death in any subject in which the cause of death is judged to have a reasonable possibility of relatedness to the study intervention by the investigator.
   * >20% of the enrolled subjects experience clinically significant grade 3/4 AEs or confirmed grade 3/4 laboratory abnormalities considered by the investigator to have a reasonable possibility of relatedness to the study intervention.
   * Investigators will inform the ethics committee with all details of each patient included in the study .investigators will stop the study once ethical committee informed us to stop according to committee rules.
3. BENEFITS:

   Direct benefits for patients:
   * Remission of patients' autoimmune disorder directly by infused T regulatory cells. It will be checked by detecting disease severity and activity scores and follow up investigations.
   * Adoptive T cell transfer will give a chance for refractory autoimmune disease patients for control.

   Indirect benefits
   * Adoptive T reg cell transfer allows for autoimmune disease control without global suppressive of the immune system by immunosuppressive medications.
   * Treg transfer helps in autoimmune disease control and protect patients from chronic progressive morbidity and mortality.
   * Being not expensive in comparison to other treatment options makes it achieve affordability.
   * Adoptive Treg cells are autologous with less susceptibility to adverse events (achieving safety).
   * Being a great hope for patients with advanced autoimmune diseases who are refractory to conventional available treatment, and could not reach other unavailable treatment options listed in the international guidelines. In such advanced stages, adoptive T cells can offer more improvement in the patients' quality of life, tolerability, and compliance.
   * Positive results of this study highly contributes to the welfare of Egyptian citizens
   * Help a significant subset of patients with advanced autoimmune diseases with an affordable treatment will reduce the financial burden on the Egyptian government.
   * Offering such innovative line of treatment for autoimmune patients will raise the rank of the country universities among their counterparts all over the world
   * Moving wide steps in this field could drive us to the station of using adoptive T cell transfer to prevent autoimmune diseases before completing the criteria for disease diagnosis, or even conserve central tolerance and prevent the occurrence of these diseases. This will be considered a giant step in the autoimmune diseases field.
4. PRIVACY AND CONFIDENTIALITY investigators will deal in complete confidentiality, and no one has right to read our patient medical information except the main researcher. After the research is complete, our patient's research results and also further information regarding our patient's health status will be informed .Individuals' confidentiality will be maintained in all published and written data resulting from the study.
5. Alternatives to participating:

   Patient has the right to refuse or withdraw from the study at any time. In case of refusing to participate in this research, the patient will be followed up and will receive his treatment as planned. Patient can stop participation in the study at any time without plenty or loss of patients medical care.
6. CONSENT PROCEDURES:

Rheumatology and endocrinology investigators (ASU) hospitals will obtain a written consent. The consent will be conducted to the patient by the mentioned investigator during the first visit. Literate individuals will be left to read the consent followed by its explanation by the mentioned investigator, while illiterate individuals will have the consent read and explained to them as well.

ELIGIBILITY:
Group 1: refractory lupus nephritis

Inclusion Criteria:

1. Patients diagnosed as refractory lupus nephritis .
2. Hemoglobin level> or equal 11g/dl before withdrawal of blood from patient to isolate T reg cells.
3. Written informed consent from every patient before participation.

Exclusion Criteria:

1. Diabetes mellitus
2. End-stage renal disease.
3. Pregnant and lactation.
4. Patients on treatment by high-dose glucocorticoids more than 20 mg/day at the time of enrollment.
5. Patients having psychiatric or neurological disease interfere with getting informed consent.
6. Patients having fever, local or systemic infection at time of administration of adoptive T reg cells.
7. Age less than or equal 18 years old.
8. Patients with other autoimmune disease.
9. Vitamin D deficient patients

Group 2: type 1 diabetes Meletus

Inclusion criteria:

1. Documented Autoimmune type 1 diabetes Meletus (TID) with disease duration ≤ 1 year, Anti GAD antibodies will be measured to all recruited patients to document autoimmunity.
2. Age ≥ 18 years old.
3. Fasting plasma C-peptide levels >0.4 ng/mL.
4. Patients on basal-bolus therapy
5. HbA1c % ≤ 8%
6. Hemoglobin level> or equal 11g/dl before withdrawal of blood from patient to isolate T reg cells.
7. Written informed consent from every patient before participation.

Exclusion criteria:

1. Patients having, fever, local or systemic infection at time of infusion of adoptive T reg cells.
2. Patient having coronary heart disease
3. End-stage renal disease
4. Pregnant and lactating patients
5. Patients having psychiatric or neurological disease interfere with getting informed consent.
6. Patients having other autoimmune disease other than TID.
7. Vitamin D deficient Patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Safety of the adoptive T regs transfer | 4 weeks
  percentage of patients who developed toxic adverse events
Efficacy of the adoptive T regs transfer | 44 weeks
  Serum detection of INF-gama,TNF-alpha,IL1,IL2,TGF-beta,IL-10,IL-17

SECONDARY OUTCOMES:
Prevention or stop progression to organ failure | 44 weeks
  percentage of patients who developed renal failure in first group and who increased the dose of insulin in the second group.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, faculty of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided